CLINICAL TRIAL: NCT05437185
Title: The Transcranial Direct Current Stimulation Treatment of Tinnitus and Its Psychiatric Comorbidities
Brief Title: Long-term tDCS Tinnitus Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Jozef Buday, Head of the Neurostimulation Center; Assistant Professor, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 531/19 S-IV
Record Dates: First submitted 2022-06-20; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Tinnitus
Keywords: tDCS; tinnitus; anxiety; depression; neurostimulation
MeSH Terms: conditions — Tinnitus; Anxiety Disorders; Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants were randomly allocated either to the active or sham (placebo) group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants were distributed between 2 arms using an aperiodic, nondeterministic, atmospheric random noise randomization algorithm. The stimulation type was unblinded upon completing all the follow-ups or dropping out. The blinding was ensured by a dedicated team member with no direct access to the participants or their data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active group (Active Comparator): The investigators aimed for six sessions of anodal stimulation over the right DLPFC (F4 in 10-20 EEG system) with cathode above the left DLPFC (F3) using HDCstim by Newronika S.r.l., Italy. The therapy was administered over two weeks (Mon, Wed, Fri) to ensure a washout period of 48 to 72 hours between applications. The current of 1.5 mA was delivered via silicone electrodes inserted into saline (0.9%) filled cellulose sponges, both 5x5cm (Current Density of 0.6 A/m2), for 20 minutes with 20 seconds of both ramp-up and ramp-down. An International 10-20 EEG system was used to determine the stimulation location, and dedicated EEG caps were used to ensure consistency between applications.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham group (Placebo Comparator): The sham (placebo) was administered using the same devices with a preprogrammed sham protocol (using HDCprog by Newronika S.r.l., Italy) of 20 minutes to be virtually indistinguishable from the active stimulation.
  Interventions: Device: Sham Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Transcranial Direct Current Stimulation (tDCS) is a non-invasive neuromodulatory method utilizing weak electrical currents to elicit short and long-term central nervous system changes.
  Arms: Active group
Device: Sham Transcranial Direct Current Stimulation — The sham was administered using the same tDCS devices as in the active group with a preprogrammed sham protocol of 20 minutes to be virtually indistinguishable from the active stimulation.
  Arms: Sham group

SUMMARY:
The study was designed to evaluate a therapeutic effect of tDCS in the treatment of tinnitus and its comorbidities (anxiety, depresion) and to evaluate the associated quality of life.

In the randomized, double-blinded, sham-controlled trial, 39 participants (active n=19, sham n=20) underwent bilateral dorsolateral prefrontal cortex (DLPFC) tDCS (anode over right DLPFC, cathode left DLPFC, current of 1.5 mA, 20 minutes, 6 sessions in 2 weeks). Tinnitus Functional Index (TFI), Iowa Tinnitus Handicap Questionnaire (ITHQ), Beck Anxiety Inventory (BAI), Zung Self-Rating Depression Scale (SDS), and WHO-Quality of Life-BREF were employed in 4 evaluation points, including the follow-ups of 6 weeks and six months.

DETAILED DESCRIPTION:
A prospective, randomized, double-blinded, placebo-controlled, two-arm trial was conducted at the Department of Psychiatry, General University Hospital in Prague, Czechia. The research was conducted in accordance with the Declaration of Helsinki and was approved by the Ethics Committee of General University Hospital in Prague, Czechia, in 2019 under the reference number 531/19 S-IV.

Participants were recruited through the recruitment campaign of the Department of Psychiatry, which was supported by outpatient services of several neurological, psychiatric, internal, and otorhinolaryngological departments in several university hospitals around Prague. All participants were required to sign written consent with the trial, anonymized data, the European Union General Data Protection Regulation (GDPR), and were fully informed about the trial's goals, risks, and requirements. Participation was not associated with any financial reward.

The participation was offered to persons at least 18 years of age (on the day of signing the consent) with a history of tinnitus lasting at least six months. The investigators excluded persons contraindicated to tDCS - such as those with epilepsy, intracranial masses or metallic objects, pregnancy, and heart conditions. The investigators also excluded persons with a history of alcohol and drug abuse, persons unwilling to sign the informed consent or persons who underwent any other tinnitus therapy in the last six months. The investigators intended to discontinue the treatment in any participant developing any severe adverse effect (significant exacerbation of tinnitus, epileptic seizure, severe headache, or any adverse effect deemed severe enough by the participants) and in participants noncompliant or unwilling to participate further with the trial and its follow-ups. The investigators required the participants not to alter their medication at least six months before the trial if any was used.

ELIGIBILITY:
Inclusion Criteria:

* Nonpulsatile tinnitus for at least 6 months
* 18 and more years of age

Exclusion Criteria:

* Pregnancy
* Unstable cardiovascular condition
* History of seizures
* Intracranial masses
* Intracranial metalic objects
* History of alcohol or drug abuse
* Unwillingness to sign the informed consent
* Inability to pass the follow-up
* Unstable medication for at least 6 months prior to the enrollment
* Other stimulation method for at least 6 months prior to the enrollmment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Tinnitus Functional Index (TFI) at T1 (baseline) | The measurement was established as a baseline prior to the stimulation series. (at T1)
  A questionaire evaluating 8 subdomains of tinnitus. A total minimal score=0, maximum score=250. Higher score means generally more severe form of tinnitus.
Changes in Tinnitus Functional Index (TFI) at T2 | Measured at T2 (after the 6th stimulation, 2 weeks since T1)
  Changes compared to the baseline (T2-T1) were calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement.
Changes in Tinnitus Functional Index (TFI) at T3 | Measured at T3 (6 weeks since T1)
  Changes compared to the baseline (T3-T1) were calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement.
Changes in Tinnitus Functional Index (TFI) at T4 | Measured at T4 (6 months since T1)
  Changes compared to the baseline (T4-T1) were calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement.
Iowa Tinnitus Handicap Questionnaire version 1 (ITHQ) at T1 (baseline) | The measurement was established as a baseline prior to the stimulation series. (at T1)
  A questionnaire evaluating 3 subdomains of tinnitus and its handicap. A total minimal score=0 %, maximum score=100%. Higher score means generally more severe form of tinnitus.
Changes in Iowa Tinnitus Handicap Questionnaire version 1 (ITHQ) at T2 | Measured at T2 (after the 6th stimulation, 2 weeks since T1)
  Changes compared to the baseline (T2-T1) were calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement.
Changes in Iowa Tinnitus Handicap Questionnaire version 1 (ITHQ) at T3 | Measured at T3 (6 weeks since T1)
  Changes compared to the baseline (T3-T1) were calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement.
Changes in Iowa Tinnitus Handicap Questionnaire version 1 (ITHQ) at T4 | Measured at T4 (6 months since T1)
  Changes compared to the baseline (T4-T1) were calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement.
Beck Anxiety Inventory (BAI) at T1 (baseline) | The measurement was established as a baseline prior to the stimulation series. (at T1)
  A standardized questionaire to evaluate the symptoms of anxiety. Minimum=0 points, maximum=63 points. A higher score means generally more severe anxiety.
Changes in Beck Anxiety Inventory (BAI) at T2 | Measured at T2 (after the 6th stimulation, 2 weeks since T1)
  Changes compared to the baseline (T2-T1) were calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement.
Changes in Beck Anxiety Inventory (BAI) at T3 | Measured at T3 (6 weeks since T1)
  Changes compared to the baseline (T3-T1) were calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement.
Changes in Beck Anxiety Inventory (BAI) at T4 | Measured at T4 (6 months since T1)
  Changes compared to the baseline (T4-T1) were calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement.
Zung Self-Rating Depression Scale (SDS) at T1 (baseline) | The measurement was established as a baseline prior to the stimulation series. (at T1)
  A standardized questionaire focusing on symptoms of depression. The scale calculates SDS index from the raw data - minimal SDS index=25 points; maximal SDS index=100 points. Higher SDS index means generally more severe depression.
Changes in Zung Self-Rating Depression Scale (SDS) at T2 | Measured at T2 (after the 6th stimulation, 2 weeks since T1)
  Changes compared to the baseline (T2-T1) were calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement.
Changes in Zung Self-Rating Depression Scale (SDS) at T3 | Measured at T3 (6 weeks since T1)
  Changes compared to the baseline (T3-T1) were calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement.
Changes in Zung Self-Rating Depression Scale (SDS) at T4 | Measured at T4 (6 months since T1)
  Changes compared to the baseline (T4-T1) were calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement.
The World Health Organization Quality Of Life (WHOQOL)-BREF at T1 (baseline) | The measurement was established as a baseline prior to the stimulation series. (at T1)
  An abbreviated version of WHO questionaire evaluating 4 domains of quality of life during the therapy. The outcomes are calculatefd are on a scale ranging between 0-100%. Higher scores mean generally higher perceived quality of life.
Changes in The World Health Organization Quality Of Life (WHOQOL)-BREF at 2 | Measured at T2 (after the 6th stimulation, 2 weeks since T1)
  Changes compared to the baseline (T2-T1) were calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement.
Changes in The World Health Organization Quality Of Life (WHOQOL)-BREF at 3 | Measured at T3 (6 weeks since T1)
  Changes compared to the baseline (T3-T1) were calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement.
Changes in The World Health Organization Quality Of Life (WHOQOL)-BREF at 4 | Measured at T4 (6 months since T1)
  Changes compared to the baseline (T4-T1) were calculated and further statistically compared between the groups. A negative difference to the baseline means an improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Tadeas Mares, M.D., Principal Investigator — Psychiatric Department, General University Hospital and 1st Faculty of Medicine, Prague; Martin Anders, M.D., Ph.D., Study Director — Psychiatric Department, General University Hospital and 1st Faculty of Medicine, Prague; Jozef Buday, M.D., Ph.D., Principal Investigator — Psychiatric Department, General University Hospital and 1st Faculty of Medicine, Prague
Locations (1):
- Psychiatric Department, General University Hospital and 1st Faculty of Medicine, Prague, Prague, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Yes
IPD can be shared upon request from a verified researcher.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after the final publication, indefinitely
Access Criteria: Upon individual request by a verified researcher.

REFERENCES:
- [Derived] Mares T, Albrecht J, Buday J, Podgorna G, Le TH, Magyarova E, Poshor K, Halik J, Buna J, Capek V, Kostylkova L, Klasova J, Fabian V, Anders M. Long-term effect of transcranial direct current stimulation in the treatment of chronic tinnitus: A randomized, placebo-controlled trial. Front Psychiatry. 2022 Oct 13;13:969800. doi: 10.3389/fpsyt.2022.969800. eCollection 2022. PMID 36311525